CLINICAL TRIAL: NCT05970926
Title: Normal Reference Values in Han Adults of Extremity Arterial Structure and Hemodynamics by High-frequency Ultrasound: a Multi-center Study in China
Brief Title: Normal Reference Values in Han Adults of Extremity Arterial Structure and Hemodynamics by High-frequency Ultrasound
Acronym: NOVAEA-HFUS
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: First Hospital of China Medical University (Other)
Responsible Party: Principal Investigator, Chunyan Ma, Chief of Cardiovascular Ultrasound, First Hospital of China Medical University
Other Study IDs: NOVAEA-HFUS-01
Record Dates: First submitted 2023-07-23; First posted 2023-08-01 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Healthy Volunteer; Artery Disease
Keywords: extremity arterial structure; extremity arterial blood flow; high-frequency ultrasound

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: high-frequency ultrasound — The volunteers will be given a high-frequency ultrasound examination of the extremity arteries, which is non-invasive, and the parameters of arterial structure and blood flow will be measured.

SUMMARY:
In recent years, high-frequency ultrasound, due to its higher resolution, can clearly display the superficial vascular structure and blood flow, and can detect vascular lesions early, providing a new non-invasive tool for clinical observation of the structure and blood flow of the extremity artery. The purpose of this multi-center study is to establish the normal value of high frequency ultrasound for the structure and blood flow of the extremity arteries of Chinese Han adults, and to explore the influencing factors, so as to provide a quantitative reference for the early diagnosis, degree evaluation and curative effect observation of the structure and blood flow of the extremities.

DETAILED DESCRIPTION:
The extremity artery is the peripheral blood vessel of the whole body, and it is often involved early in the diseases that are easy to damage the small vessels, such as atherosclerosis and connective tissue diseases. Early lower limb atherosclerosis mainly occurs in the dorsal foot artery, which is commonly seen in people with diabetes and long-term smoking. Connective tissue diseases such as systemic sclerosis and systemic lupus erythematosus also mainly involve small blood vessels, and vascular lesions may appear earlier than those of other specific organs such as heart and lung. Because of its shallow location, the extremity artery can be better used as a screening site for vascular diseases, and it is the window for early reaction of vascular diseases.However, the early stage of extremity artery disease is easy to be ignored, and patients often have pain and numbness of the affected limb. When the disease is severe, it can lead to ulcer not healing, and even limb gangrene and amputation, which greatly affects the quality of life and brings huge troubles and economic pressure to the patients. Therefore, early diagnosis of extremity arterial lesions is of great significance for early diagnosis of microvascular injury diseases such as atherosclerosis and connective tissue diseases, reducing the incidence of complications, and reducing the rate of amputation and mortality.

Ultrasound is a non-invasive imaging technique widely used in clinic. In recent years, with the development of ultrasound technology, the frequency of ultrasonic probes has been increasing. Because of its higher resolution, high-frequency ultrasound can clearly display the superficial vascular structure and blood flow, detect vascular lesions early, and accurately quantify the degree of stenosis, providing a new and beneficial tool for clinical observation of the structure and blood flow of the extremity artery. The purpose of this multi-center clinical study was to establish the normal value of high frequency ultrasound for the structure and blood flow of the extremities of Chinese Han adults, and to explore its influencing factors, so as to provide a quantitative reference for the early diagnosis, degree evaluation and curative effect observation of the structure and blood flow of the extremities.

ELIGIBILITY:
Inclusion Criteria:

1. Han nationality;
2. Ages 18-79;
3. Normal blood pressure (139-90/89-60mmHg);
4. Body mass index < 30 kg/m2;
5. Blood routine, fasting blood glucose, blood lipid, liver and kidney function, electrocardiogram were normal;
6. No history of cyanosis of hands and feet, cold stimulation without discomfort, no Raynaud phenomenon has occurred in all parts of the body;
7. No cardiovascular disease, diabetes, rheumatic connective tissue disease, serious liver and kidney dysfunction;
8. No history of drug use affecting cardiovascular system.

Exclusion Criteria:

1. Patients with hypertension, diabetes, hyperthyroidism, arrhythmia and other diseases;
2. Patients with systemic lupus erythematosus, polymyositis, rheumatoid arthritis and other connective tissue diseases;
3. A history of related blood diseases;
4. Have taken vasoconstrictor drugs in the past 1 month;
5. Gangrene of fingers and toes or history of trauma or surgery;
6. Have a history of handicraft, hammering, digging and other related work;
7. Have a long history of smoking and drinking;
8. Peripheral vascular disease, arterial occlusion can not detect blood flow signal;
9. Unable to cooperate with the examiner.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Chinese healthy Han adults
Sampling Method: Probability Sample
Enrollment: 540 (Estimated)
Dates: Start 2023-08-01 (Estimated); Primary Completion 2024-08-31 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Intima thickness of dorsalis pedis artery and proper palmar digital artery | 1 day
  Intima thickness reflects the changes of vascular wall structure and is used for early evaluation of arterial disease.

SECONDARY OUTCOMES:
Blood flow velocity of dorsalis pedis artery and proper palmar digital artery | 1 day
  Blood flow velocity reflects hemodynamic changes and is used for early evaluation of arterial disease.

CONTACTS AND LOCATIONS:
Overall Officials: Lixin Jiang, PHD, Principal Investigator — Shanghai Jiao Tong University School of Medicine; Xinhua Ye, PHD, Principal Investigator — The First Affiliated Hospital with Nanjing Medical University; WeiDong Ren, PHD, Principal Investigator — Shengjing Hospital; Xin Guan, PHD, Principal Investigator — Tianjin Chest Hospital; Hongning Yin, PHD, Principal Investigator — The Second Hospital of Hebei Medical University; Xiaoshan Zhang, PHD, Principal Investigator — The Affiliated Hospital of Inner Mongolia Medical University; Yuhong Zhang, PHD, Principal Investigator — The Second Affiliated Hospital of Dalian Medical University; Qingxiong Yue, PHD, Principal Investigator — Dalian Municipal Central Hospital

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol (2023-05-28): https://cdn.clinicaltrials.gov/large-docs/26/NCT05970926/Prot_000.pdf
  • Informed Consent Form (2023-05-28): https://cdn.clinicaltrials.gov/large-docs/26/NCT05970926/ICF_001.pdf